CLINICAL TRIAL: NCT04619277
Title: Impact of Drug-coated Balloon Treatment in de Novo Coronary Lesion
Status: Recruiting | Type: Observational
Sponsor: Ulsan Medical Center (Other)
Responsible Party: Principal Investigator, Eun-Seok Shin, Director, Ulsan Medical Center
Other Study IDs: USH-20-004; USH-20-004 (Registry Identifier: Ulsan Medical Center)
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Drug-coated Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (7):
- Ulsan Medical Center: Division of Cardiology, Department of Internal Medicine, Ulsan Medical Center, Ulsan, South Korea
  Interventions: Device: drug-coated balloon
- Queen Elizabeth Hospital: Cardiology Department and Clinical Research Center, Queen Elizabeth Hospital II, Kota Kinabalu, Malaysia
  Interventions: Device: drug-coated balloon
- Pecking University Shougand Hospital: Department of Cardiology, Peking University Shougang Hospital, Peking, China
  Interventions: Device: drug-coated balloon
- Ulsan University Hospital: Department of Internal Medicine, Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan, South Korea
  Interventions: Device: drug-coated balloon
- Kangwon National University School of Medicine: Department of Internal Medicine, Kangwon National University School of Medicine, Chuncheon, South Korea
  Interventions: Device: drug-coated balloon
- Korea University Guro Hospital: Cardiovascular Center, Department of Cardiology, Korea University Guro Hospital, Seoul, South Korea
  Interventions: Device: drug-coated balloon
- Korea University Ansan Hospital: Department of Cardiology, Korea University Ansan Hospital, Ansan, South Korea
  Interventions: Device: drug-coated balloon

INTERVENTIONS:
Device: drug-coated balloon — drug-coated balloon

SUMMARY:
This study is the international multicenter registry for drug-coated balloon treatment for de novo coronary lesion.

DETAILED DESCRIPTION:
There is lots of evidence that DCBs result in lower rates of restenosis, thrombosis, and better long-term outcomes when used for PCI of in-stent restenosis (ISR) compared to plain old balloon angioplasty (POBA) or additional stenting with drug-eluting stent (DES). DCB-only approach studies for de novo coronary lesion cases are scarce, but a recent registry data suggested it was a feasible and well-tolerated treatment method if the pre-dilation result is good. Therefore, the aim of this study was to evaluate the safety and efficacy in terms of angiographic and clinical outcomes of a DCB-only approach for de novo coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

- de novo coronary artery disease

Exclusion Criteria:

* unstable hemodynamics at presentation
* life expectancy <1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is a international multicenter registry study conducted at 4 centers (Queen Elizabeth Hospital II, Peking Shougang Hospital, Ulsan Medical Center, and Ulsan University Hospital) expert in patients with de novo coronary lesion who received DCB treatment.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-04-22 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events at 12 months | 12 months
  Primary endpoint is major adverse cardiac events (MACE is a composite of cardiac death, non-fatal myocardial infarction, target-vessel revascularization and major bleeding [BARC type 3 to 5]) at 12 months.
  1. Cardiac death: Any death due to proximate cardiac cause (eg, myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
  2. Target vessel Revascularization: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel.

SECONDARY OUTCOMES:
Angiographic and clinical outcomes | 12, 24, 36 months
  * MACE at 12, 24, 36 months
    * The single components of the primary endpoint after 12, 24, 36 months. Bleeding Academic Research Consortium (BARC) type 2 to 5 bleeding after 12, 24, 36 months.1 (All events will be adjudicated by an independent Critical Events Committee).
      * Possible, probable, and definite stent thrombosis defined according to the ARC criteria after 12, 24, 36 months.
        * Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation
          * Cost-effectiveness of DCB vs. DES after 12, 24, 36 months.
            * All-cause death ⑥ Stroke (ischemic and hemorrhagic)
              * Angina severity measured with Seattle Angina Questionnaires at 12, 24 months
                * Total procedure time, fluoroscopy time, contrast volume, number of stents used ⑨ DAPT duration ⑩ Periprocedural MI rate ⑪ Sex difference in MACE between DCB vs. DES ⑫ Comparison of MACE between DCB vs. DES in DM patients

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Jin Kim, Principal Investigator — IRB
Locations (1):
- Ulsan Medical Center, Ulsan, South Korea

REFERENCES:
- [Derived] Her AY, Kim S, Kang DO, Sohn CB, Kim YH, Kim B, Shin ES. Drug-Coated Balloon-Based Intervention for De Novo Acute Myocardial Infarction. Yonsei Med J. 2025 Dec;66(12):807-815. doi: 10.3349/ymj.2024.0524. PMID 41287492
- [Derived] Her AY, Kim TH, Shin ES, Kim S, Kim B, Kim YH, Choi KH, Cho YK, Lee HJ, Song YB, Nam CW, Gwon HC. Drug-Coated Balloon-Based Treatment of Left Main True Bifurcation Lesion. Catheter Cardiovasc Interv. 2025 Apr;105(5):1024-1031. doi: 10.1002/ccd.31416. Epub 2025 Jan 22. PMID 39840648
- [Derived] Her AY, Shin ES, Kim S, Kim B, Kim TH, Sohn CB, Choi BJ, Park Y, Cho JR, Jeong YH. Drug-coated balloon-based versus drug-eluting stent-only revascularization in patients with diabetes and multivessel coronary artery disease. Cardiovasc Diabetol. 2023 May 20;22(1):120. doi: 10.1186/s12933-023-01853-0. PMID 37210516
- [Derived] Shin ES, Jun EJ, Kim S, Kim B, Kim TH, Sohn CB, Her AY, Park Y, Cho JR, Jeong YH, Choi BJ. Clinical Impact of Drug-Coated Balloon-Based Percutaneous Coronary Intervention in Patients With Multivessel Coronary Artery Disease. JACC Cardiovasc Interv. 2023 Feb 13;16(3):292-299. doi: 10.1016/j.jcin.2022.10.049. Epub 2023 Jan 4. PMID 36609038
- [Derived] Jun EJ, Shin ES, Teoh EV, Bhak Y, Yuan SL, Chu CM, Garg S, Liew HB. Clinical Outcomes of Drug-Coated Balloon Treatment After Successful Revascularization of de novo Chronic Total Occlusions. Front Cardiovasc Med. 2022 Apr 13;9:821380. doi: 10.3389/fcvm.2022.821380. eCollection 2022. PMID 35498010
- [Derived] Kun L, Shin ES, Jun EJ, Bhak Y, Garg S, Kim TH, Sohn CB, Choi BJ, Hui L, Yuan SL, Zhi W, Hao J, Zhentao S, Qiang T. Sex-Related Outcomes of Successful Drug-Coated Balloon Treatment in De Novo Coronary Artery Disease. Yonsei Med J. 2021 Nov;62(11):981-989. doi: 10.3349/ymj.2021.62.11.981. PMID 34672131
- [Derived] Hui L, Shin ES, Jun EJ, Bhak Y, Garg S, Kim TH, Sohn CB, Choi BJ, Kun L, Yuan SL, Zhi W, Hao J, Zhentao S, Qiang T. Impact of Dissection after Drug-Coated Balloon Treatment of De Novo Coronary Lesions: Angiographic and Clinical Outcomes. Yonsei Med J. 2020 Dec;61(12):1004-1012. doi: 10.3349/ymj.2020.61.12.1004. PMID 33251774